CLINICAL TRIAL: NCT02273648
Title: BIOTRONIK - SaFety and Performance Registry for an All-comers Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice - III French Satellite
Brief Title: BIOTRONIK - BIOFLOW-III Registry French Satellite
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Biotronik France (Industry)
Responsible Party: Sponsor
Other Study IDs: G1401 French Satellite
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Diseases
Keywords: national; multicenter; observational registry; Orsiro Drug Eluting Stent; Stenting Treatment of coronary artery disease; coronary revascularization; PCI; STEMI; NSTEMI; Ischemia; Angina; Acute Myocardial Infarction; Small Vessels; Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris | interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro: Subjects requiring coronary revascularization with Drug Eluting Stents (DES) as well as Subjects presenting with
  1. Diabetes (all types) at least 300 subjects should be included and analyzed in this segment
  2. Small vessels (≤2.75 mm) approx. 150 subjects
  3. Chronic total occlusion (CTO) approx. 50 subjects
  4. Acute Myocardial Infarction (incl. STEMI and NSTEMI) approx. 100 subjects
  5. Multivessels approx. 250 subjects
  6. In stent restenosis approx. 100 subjects
  7. Different type of DAPT interruption : <3 months, between 3 and 6 months, after 6 months approx. 300 subjects subjects who stopped <3 months
  Interventions: Device: Drug Eluting Stent (DES)

INTERVENTIONS:
Device: Drug Eluting Stent (DES) — Percutaneous Coronary Intervention

SUMMARY:
For the majority of Coronary Artery Disease (CAD) treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedure success. However, the medium to long-term complications range from rather immediate elastic coil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30 to 50%. Such rates of recurrence have serious economic consequences. Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in De Novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20 to 40% of cases, necessitating repeat procedures.

The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilized on the stent surface or released from a polymer matrix), which inhibits neointimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in better safety profile as compared to BMS with systemic drug administration. These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease.

Therefore this observational registry has been designed for the clinical evaluation of the ORSIRO LESS requiring coronary revascularization with DES. It is designed to investigate and collect clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in an all-comers patient population in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease
* Subject has signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow up assessments
* Subject is ≥ 18 years of age

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Pregnancy
* Known intolerance to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI, stainless steel, Sirolimus or contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects requiring coronary revascularization with Drug Eluting Stents (DES)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG) and clinically driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
TLF | 6, 24, 36, 48 and 60 months
  Defined as the composite of Cardiac death, Target vessel Q-wave or non-Q wave Myocardial Infarction (MI) (i.e., Q-wave MI that cannot be attributed to a non-target vessel), clinically driven Target Lesion Revascularization (TLR) and Emergent Coronary Artery Bypass Grafting (CABG).
Target Vessel Revascularization (TVR) | 6, 12, 24, 36, 48 and 60 months
  Any repeat revascularization of the target vessel. (Vascular bypass or angioplasty)
Target Lesion Revascularization (TLR) | 6, 12, 24, 36, 48 and 60 months
  Target Lesion Revascularization (Vascular bypass or angioplasty)
Stent Thrombosis | 6, 12, 24, 36, 48 and 60 months
  Definite, Probable and Possible Stent Thrombosis
Clinical Device Success | up to 1 day
  Successful delivery and deployment of the investigational stent (s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation and without use of a device outside the assigned treatment strategy.
Clinical Procedural Success | up to seven days
  Successful delivery and deployment of the investigational stent(s) at the intended target lesion (this includes successful delivery and deployment of multiple overlapping stents, if applicable) and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% of the target lesion as observed by visual estimate without using any adjunctive device* without the occurrence of ischemia-driven major adverse cardiac event (ID-MACE) during the hospital stay to a maximum of the first seven days post index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CANOT, Study Director — Biotronik France
Locations (50):
- France (50):
  - CH d'Aix en Provence, Aix-en-Provence
  - Clinique de l'Europe, Amiens
  - Centre Hospitalier d'Antibes, Antibes
  - Clinique Rhône Durance, Avignon
  - Hopital Henri Duffaut, Avignon
  - Centre Hospitalier de Bastia, Bastia
  - Clinique la fourcade, Bayonne
  - Clinique St Augustin, Service Cardiologie Interventionnelle, Bordeaux
  - Clinique Convert, Cardiologie Interventionnelle, Bourg-en-Bresse
  - Clinique Keraudren, Brest
  - HP St Martin, Service de Cardiologie, Caen
  - CHU de Clermont Ferrand, Hôpital Gabriel Montpied, Clermont-Ferrand
  - CH Sud Francilien, Corbeil
  - Clinique Louis Pasteur, Essey-lès-Nancy
  - CHU Fort de France, Fort-de-France
  - Groupe Hospitalier Mutualiste, Grenoble
  - CHU Point-à-Pitre, La Guadeloupe
  - Centre Hospitalier de la Roche-sur-Yon, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH de Versailles, Le Chesnay
  - Hôpital Louis Pasteur, Le Coudray
  - Hôpital privé de l'Estuaire, Le Havre
  - CHRU de Lille, Lille
  - Lyon Saint Joseph Saint Luc, Lyon
  - CHU de la Timone, Marseille
  - Hôpital Nord de Marseille, Service de Cardiologie, Marseille
  - Clinique les Fontaines, Melun
  - Centre Hospitalier Annecy, Metz-Tessy
  - Clinique Pont de Chaume, Montauban
  - Montpellier le Millenaire, Montpellier
  - Clinique du Diaconat Fonderie, Mulhouse
  - CHU de Nantes, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU Nimes, Nîmes
  - Polyclinique les Fleurs, Ollioules
  - Centre Hospitalier de Pau, Pau
  - Hôpital Privé St Martin, Pessac
  - Hôpital privé Claude Galien, Quincy
  - Clinique Saint Hilaire, Rouen
  - Centre Hospitalier St Brieuc, Saint-Brieuc
  - Centre Cardiologique du Nord (CCN), Saint-Denis
  - CHU Reunion, Saint-Denis
  - Clinique Ste Clotilde, Sainte-Clotilde
  - Clinique de l'Orangerie, Strasbourg
  - Nouvel Hôpital Civil, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - Clinique St Gatien, Tours
  - Clinique St Joseph, Trélazé
  - CH de Valence, Valence
  - CHIV de Villeneuve St Georges, Villeneuve-Saint-Georges